CLINICAL TRIAL: NCT01901016
Title: Relaxation, Depressive Symptoms, Quality of Life, Immunological and Virological Status o in People Living With HIV: a Pilot Study
Brief Title: Relaxation, Depressive Symptoms, Quality of Life in People Living With HIV: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: RRISIQ (Unknown); Laval University (Other)
Responsible Party: Principal Investigator, Pilar Ramirez-Garcia, RN, PhD, Assistant Professor, Faculty of nursing & Researcher at CHUM research centre, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RELHIV-13
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2018-05

CONDITIONS: HIV; Depressive Symptoms
Keywords: HIV; depressive symptoms; quality of life; relaxation; viral load; CD4+ T cell count
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Jacobson progressive muscular relaxation (Experimental): Jacobson progressive muscular relaxation
  Interventions: Behavioral: Jacobson progressive muscular relaxation
- Schultz's autogenic training (Experimental): Schultz's autogenic training
  Interventions: Behavioral: Schultz's autogenic training
- control (No Intervention): The CG continued to receive their standard care. After data collection at the six-month follow-up, the CG participants were invited to attend one of two relaxation interventions.

INTERVENTIONS:
Behavioral: Jacobson progressive muscular relaxation — PMR involves learning to identify the tension in specific muscle groups by tightening and relaxing each muscle group. It includes three different exercises: 1) contraction-relaxation of 12 large muscle groups in the arms, legs, and trunk; 2) identification and relaxation of tensions without the need for movement or contractions; and 3) contraction-relaxation of 12 small muscle groups in the neck, eyes, and mouth
  Arms: Jacobson progressive muscular relaxation
Behavioral: Schultz's autogenic training — AT is a relaxation technique that is based on body attitude, reduction of exterior stimulation, inner concentration, and mental repetition of verbal formulas [28]. These formulas are organized into six exercises: 1) heaviness; 2) warmth; 3) calm and regular heart function; 4) self-regulation of respiration; 5) warmth in the upper abdominal area; and 6) agreeable cooling of the forehead.
  Arms: Schultz's autogenic training

SUMMARY:
Progressive muscle relaxation (PMR) and autogenic training (AT) are effective relaxation techniques to reduce depressive symptoms. However, no studies on their effectiveness have been conducted among people living with HIV and depressive symptoms. The primary aim of this pilot study was to assess the feasibility and acceptability of PMR and AT interventions among people living with HIV who have depressive symptoms. A secondary aim was to assess the potential effectiveness of these interventions on depressive symptoms and quality of life.

DETAILED DESCRIPTION:
This study was a three-arm pilot randomized control trial with mixed methods. Participants were randomized to PMR, AT, or control group (CG), with four assessments (baseline, one-, three-, and six-month). The PMR and AT interventions consisted of six one-hour sessions of individual training over 12 weeks and home practice. Recruitment, attrition, and completion rates were calculated. Depressive symptoms and quality of life were assessed at all times. Participants' perceptions of the interventions were collected in semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* HIV diagnosis of at least two years
* Depressive symptoms between 5 and 14 in the PHQ-9 scale
* Untreated with antidepressants or psychotherapy
* Able to speak and understand French

Exclusion Criteria:

* Started antiretroviral treatment within the last 6 months
* Start or already receiving Interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms measured with Personal Health Questionnaire (PHQ-9) assessed at 3 months | baseline and 3 months
  Depressive symptoms at 3 months will be measured with Personal Health Questionnaire (PHQ-9)
Change from baseline in depressive symptoms measured with Personal Health Questionnaire (PHQ-9) assessed at 6 months | baseline and 6 months
  Depressive symptoms at 6 months will be measured with Personal Health Questionnaire (PHQ-9)
Change from baseline in depressive symptoms measured with Personal Health Questionnaire (PHQ-9)assessed at 1 month | baseline and 1 month
  Depressive symptoms at 1 month will be measured with Personal Health Questionnaire (PHQ-9)

SECONDARY OUTCOMES:
Change from baseline in quality of life measured with (MOS-HIV) Medical Outcome Study-HIV assessed at 6 months | baseline and 6 months
  Quality of life at 6 months will be measured with MOS-HIV) Medical Outcome Study-HIV
Change from baseline in quality of life measured with MOS-HIV) Medical Outcome Study-HIV assessed at 3 months | baseline and 3 months
  Quality of life at 3 months will be measured with MOS-HIV) Medical Outcome Study-HIV

OTHER OUTCOMES:
Change from baseline in viral load assessed at 6 months | baseline and 6 months
  Change from baseline in viral load assessed at 6 months
Change from baseline in CD4+ T cells count at 6 months | baseline and 6 months
  Change from baseline in CD4+ T cells count at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Ramirez Garcia, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Research center CHUM, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Ramirez Garcia MP, Leclerc-Loiselle J, Cote J, Brouillette MJ, Thomas R. Effect of autogenic training on quality of life and symptoms in people living with HIV: A mixed method randomized controlled trial. Complement Ther Clin Pract. 2023 Feb;50:101716. doi: 10.1016/j.ctcp.2022.101716. Epub 2022 Dec 13. PMID 36528982
- [Derived] Ramirez-Garcia MP, Leclerc-Loiselle J, Gagnon MP, Cote J, Brouillette MJ, Thomas R. A mixed-method randomized feasibility trial evaluating progressive muscle relaxation or autogenic training on depressive symptoms and quality of life in people living with human immunodeficiency virus (HIV) who have depressive symptoms. J Complement Integr Med. 2020 Jul 3;18(1):165-174. doi: 10.1515/jcim-2019-0167. PMID 32621729